CLINICAL TRIAL: NCT02582489
Title: Prospective, Randomized, Double-blind Clinical Trial to Investigate the Efficacy of Autologous Bone Marrow Aspirate Concentrate Post-Meniscectomy
Brief Title: Autologous Bone Marrow Aspirate Concentrate in Patients Undergoing Meniscectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15090903
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis Post-meniscectomy
Keywords: Mesenchymal stem cells; Bone marrow aspirate concentrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Meniscectomy with Bone Marrow Aspirate Concentrate (BMAC) (Experimental): Subjects will undergo the scheduled meniscectomy procedure. Following the procedure the investigator will make a small incision and create the marrow access channel in the proximal tibia. The experimental group will then have bone marrow harvested and BMAC will be prepared using a BMAC harvesting system. The automated centrifuge system rapidly concentrates cellular contents and growth factors in bone marrow aspirate using flow cytometry. The BMAC will be injected intra-articularly.
  Interventions: Biological: Bone Marrow Aspirate Concentrate; Procedure: Standard Meniscectomy
- Meniscectomy with Placebo (Placebo Comparator): Subjects will undergo the same meniscectomy procedure and will also have an incision and marrow access channel made in the proximal tibia, however no bone marrow will be harvested. The control group will have a placebo injection of saline into the affected knee.
  Interventions: Procedure: Standard Meniscectomy

INTERVENTIONS:
Biological: Bone Marrow Aspirate Concentrate — Subjects undergoing autologous bone marrow aspirate concentrate will receive an intra-articular injection into the affected knee.
  Arms: Meniscectomy with Bone Marrow Aspirate Concentrate (BMAC)
Procedure: Standard Meniscectomy — All subjects will undergo either a partial or complete meniscectomy to treat the torn meniscus.

SUMMARY:
The proposed research study aims to evaluate the effects of autologous bone marrow aspirate concentrate (BMAC) on the development and progression of osteoarthritis (OA) in patients undergoing meniscectomy. This prospective, randomized, double-blind clinical trial will compare patient-reported outcomes, specifically IKDC scores between patients who receive BMAC post-meniscectomy and those who receive a saline control injection. The study will also compare physical examination, MRI, radiographs, and synovial fluid analysis. Our hypothesis is that those who receive the autologous BMAC injection after the procedure will have better outcomes than those who do not.

DETAILED DESCRIPTION:
Recent studies have demonstrated both the safety of BMAC intra-articular injection and improvements in subjective, patient reported outcomes in patients with existing knee OA. Unfortunately these studies were largely uncontrolled, underpowered, and/or retrospective in nature. Additionally, a recent prospective, randomized clinical study of allograft mesenchymal stem cells (MSCs) injected at a separate time point post surgical intervention has highlighted the ability of MSCs to increase meniscal volume and improve knee pain following injection.

This will be the first study to examine the effects of autograft BMAC intra-articular injection in a single-stage procedure and in a prospective, randomized, double-blind fashion. The results of this study, if the null hypothesis is rejected, will have far-reaching implications for the standard of care in meniscal treatment and on OA progression in the knee. Additionally, if the results of this study are favorable in reduction of OA progression this study will change the surgical approach to all axial, synovial joints including the shoulder, elbow, wrist, hip, and ankle.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than 18 years old
* Written informed consent is obtained
* Subject is determined to have a symptomatic meniscal tear requiring a meniscectomy
* Meniscal pathology is confirmed through MRI and arthroscopically
* Subject agrees to all follow-up evaluations
* Osteoarthritis Kellen-Lawrence grade 1-3 on flexion PA and extension AP views

Exclusion Criteria:

* Any subject lacking decisional capability
* Unwillingness to participate in the necessary follow-up
* Subject is pregnant or may become pregnant
* History of diabetes mellitus
* History of rheumatoid arthritis or other autoimmune disorder
* History of solid organ or hematologic transplantation
* Diagnosis of a non-basal cell malignancy within the preceding 5 years
* Infection requiring antibiotic treatment within the preceding 3 months
* Osteoarthritis Kellen-Lawrence grade 4 on flexion posterior-anterior (PA) or extension anteroposterior (AP) views
* Prior surgery on the index meniscus
* Concomitant surgery such as ligament surgery or cartilage repair or restoration
* Infection
* Prior cortisone/viscosupplementation/ (platelet rich plasma) PRP injection within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score | One Year
  The primary outcome measure will be the IKDC score at one year follow-up

SECONDARY OUTCOMES:
Patient reported outcomes throughout follow-up period | 7-10 days, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Patient reported outcomes will include change in scores from preoperative to Postoperative Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Synovial fluid analysis | 2 weeks, 6 weeks
  To investigate any changes in synovial fluid markers of osteoarthritis.
Radiographic analysis | 1 year, 2 years
  The degree of OA will be examined in all patients preoperatively and at subsequent follow-up visits at 1 and 2 years.
Patient reported outcomes throughout follow-up period (VAS) | 7-10 days, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Visual Analog Score (VAS)
Patient reported outcomes throughout follow-up period (IKDC) | 7-10 days, 6 weeks, 3 months, 6 months, 1 year, 2 years
  International Knee Documentation Committee form (IKDC)
Patient reported outcomes throughout follow-up period (KOOS) | 7-10 days, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Knee injury and Osteoarthritis Outcome Score (KOOS)
Patient reported outcomes throughout follow-up period (SF-12) | 7-10 days, 6 weeks, 3 months, 6 months, 1 year, 2 years
  (Short Form Health Survey) SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Cole, MD, MBA, Principal Investigator — Midwest Orthopaedics at Rush
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Fortier LA, Potter HG, Rickey EJ, Schnabel LV, Foo LF, Chong LR, Stokol T, Cheetham J, Nixon AJ. Concentrated bone marrow aspirate improves full-thickness cartilage repair compared with microfracture in the equine model. J Bone Joint Surg Am. 2010 Aug 18;92(10):1927-37. doi: 10.2106/JBJS.I.01284. PMID 20720135
- [Background] Gobbi A, Karnatzikos G, Scotti C, Mahajan V, Mazzucco L, Grigolo B. One-Step Cartilage Repair with Bone Marrow Aspirate Concentrated Cells and Collagen Matrix in Full-Thickness Knee Cartilage Lesions: Results at 2-Year Follow-up. Cartilage. 2011 Jul;2(3):286-99. doi: 10.1177/1947603510392023. PMID 26069587
- [Background] Enea D, Cecconi S, Calcagno S, Busilacchi A, Manzotti S, Gigante A. One-step cartilage repair in the knee: collagen-covered microfracture and autologous bone marrow concentrate. A pilot study. Knee. 2015 Jan;22(1):30-5. doi: 10.1016/j.knee.2014.10.003. Epub 2014 Nov 20. PMID 25480381
- [Background] Kim JD, Lee GW, Jung GH, Kim CK, Kim T, Park JH, Cha SS, You YB. Clinical outcome of autologous bone marrow aspirates concentrate (BMAC) injection in degenerative arthritis of the knee. Eur J Orthop Surg Traumatol. 2014 Dec;24(8):1505-11. doi: 10.1007/s00590-013-1393-9. Epub 2014 Jan 8. PMID 24398701
- [Background] Centeno C, Pitts J, Al-Sayegh H, Freeman M. Efficacy of autologous bone marrow concentrate for knee osteoarthritis with and without adipose graft. Biomed Res Int. 2014;2014:370621. doi: 10.1155/2014/370621. Epub 2014 Sep 7. PMID 25276781
- [Background] Vangsness CT Jr, Farr J 2nd, Boyd J, Dellaero DT, Mills CR, LeRoux-Williams M. Adult human mesenchymal stem cells delivered via intra-articular injection to the knee following partial medial meniscectomy: a randomized, double-blind, controlled study. J Bone Joint Surg Am. 2014 Jan 15;96(2):90-8. doi: 10.2106/JBJS.M.00058. PMID 24430407
- [Derived] Yanke AB, Yazdi AA, Weissman AC, Wagner KR, Meeker ZD, Condron NB, Darwish RY, Drager J, Danilkowicz RM, Forsythe B, Verma NN, Cole BJ. A Prospective, Randomized, Double-Blind Clinical Trial to Investigate the Efficacy of Autologous Bone Marrow Aspirate Concentrate During Arthroscopic Meniscectomy in Patients With Early Knee Osteoarthritis. Am J Sports Med. 2024 Oct;52(12):2963-2971. doi: 10.1177/03635465241275647. Epub 2024 Sep 15. PMID 39279266